CLINICAL TRIAL: NCT05611892
Title: Phase 1 Biodistribution and Pathophysiology Study of 18F-Fluorodeoxysorbitol (18F-FDS)
Brief Title: Biodistribution and Pathophysiology Study of 18F-Fluorodeoxysorbitol (18F-FDS) in Diseased Patients
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00097331
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Enterobacterial Infections; Oncologic Disease; Inflammatory Disease; Invasive Fungal Infections
Keywords: PET/CT; 18F-FDS
MeSH Terms: conditions — Enterobacteriaceae Infections; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18F-FDS PET/CT: a single intravenous dose of 18F-FDS followed by PET/CT scan.
  Interventions: Combination Product: 18F-FDS PET/CT

INTERVENTIONS:
Combination Product: 18F-FDS PET/CT — 20 millicurie (mCi) of 18F-FDS in adult patient age group and 2.5 mCi in children (age 12-18 years old) followed by a PET/CT scan.

SUMMARY:
In this study, the investigators will assess the hypothesis that this new positron emission tomography (PET) radiopharmaceutical, 18F-Fluorodeoxysorbitol (18F-FDS), will specifically localize at sites of Gram-negative bacterial due to Enterobacterales and invasive mold infections (e.g. invasive aspergillosis/mucormycosis).

ELIGIBILITY:
Inclusion criteria:

Subjects may be enrolled into this protocol only if all of the following criteria are met:

1. Male or female >12 years of age at the time of consent and imaging. No healthy adolescent subjects will be enrolled in the study.
2. For inpatients, determined by the attending of record to be stable to participate in the study (will be documented in the research records).
3. For invasive mold infections - signs and symptoms clinically compatible with PROVEN or PROBABLE active invasive mold disease as determined by The European Organization for Research and Treatment of Cancer and the Mycoses Study Group Education and Research Consortium (EORTC/MSGERC) consensus definitions:

   PROVEN disease: Biopsy or needle aspiration positive for organism (i.e., hyphae, yeast cells, etc.) on microscopic examination or culture, OR nucleic acid diagnosis (i.e., PCR), OR blood culture.

   PROBABLE disease: POSITIVE galactomannan EIA based on clinically acceptable cutoff as follows:
   1. Single serum or plasma >=1.0
   2. BAL >=1.0
   3. Single serum or plasma >=0.7 and BAL fluid >=0.8 CSF >1
4. For Enterobacterales infections - clinically compatible illness plus one or more of the following:

   1. Confirmed (microbiologically, molecular or serological testing) diagnosis of infection at anybody site OR
   2. clinical and imaging evidence of suspected infection in any body site with confirmation (microbiologically, molecular or serological testing) anticipated within 72 hours of imaging.
5. For non-infectious control patients: Subjects with confirmed inflammatory (rheumatoid arthritis, idiopathic pulmonary fibrosis, etc) or oncologic (e.g. localized or metastatic tumors) disease and clinically determined not to have infection.
6. Subject is judged by the investigator to have the initiative and means to be compliant with the protocol.
7. Subjects or their legal representatives must have the ability to read, understand and provide written informed consent for the initiation of any study related procedures. Adults lacking capacity will not be enrolled in this study.

Exclusion criteria:

Within 28 or fewer days prior to imaging, a complete blood count with differential, blood comprehensive metabolic panel will be performed. Subjects will be excluded from enrollment if any of the following apply:

1. Reported pregnancy or pregnancy as determined by positive or indeterminate serum human chorionic gonadotrophin (hCG) at screening and positive urine hCG prior to radiopharmaceutical dosing.
2. Lactating females
3. History of significant renal or hepatobiliary diseases (Serum creatinine > 3 times the upper limit of normal or Total bilirubin > 3 times the upper limit of normal or Liver Transaminases > 5 times the upper limit of normal)
4. Inadequate venous access
5. Administered a radioisotope within 5 physical half-lives as part of a research study prior to study enrollment
6. Subject has been treated with an investigational drug / biologic / therapeutic device within 30 days prior to study radiotracer administration
7. Determined to have prior (external) radiation exposure from research studies which will exceed RDRC annual radiation exposure limit of 5 rems.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and female members of all races and ethnic groups are eligible for this trial and encouraged to participate
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Biodistribution of 18F-FDS in diseased subjects | Up to 3 hours
  Reconstruction of the PET data will be performed by means of iterative reconstruction (IR) by the ordered subset-expectation-maximization method with CT attenuation correction. Volumes of interest will be drawn on fused PET and CT images across different body compartments and comparison.
Pathophysiology of 18F-FDS in diseased subjects | Up to 3 hours
  Reconstruction of the PET data will be performed by means of iterative reconstruction by the ordered subset-expectation-maximization method with CT attenuation correction. Volumes of interest will be drawn on fused PET and CT images. Data will be presented as target-to-nontarget ratio (TNT), defined as the ratio of the PET signal at the sites of pathology to the unaffected sites of the same tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Jain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States